CLINICAL TRIAL: NCT03080181
Title: Adipokine Profile in Patients With Cushing's Disease on Pasireotide Treatment: Correlation With Disease Activity, Insulin Sensitivity and Secretion Parameters
Brief Title: Adipokine Profile in Patients With Cushing's Disease on Pasireotide Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Carla Giordano, Professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pasireotide-CD
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pasireotide (Experimental): Pasireotide was administered in a 12 months period
  Interventions: Drug: Pasireotide 0.6 MG/ML

INTERVENTIONS:
Drug: Pasireotide 0.6 MG/ML — The aim of the study was to evaluate the effect of pasireotide on β -cell and adipose function in patients with Cushing's disease (CD).

SUMMARY:
Background: Pasireotide treatment is strictly associated with glucose metabolism impairment. The aim of the study was to evaluate the effect of pasireotide on β -cell and adipose function in patients with Cushing's disease (CD).

Methods: Clinical and hormonal parameters, insulin secretion, evaluated by homostasis model assessment (HOMA-β) and by the area under the curve (AUC2h) of C-peptide during a mixed meal tolerance test and insulin sensitivity, evaluated by the euglycemic hyperinsulinemic clamp, were evaluated in 12 patients with active CD before and after 12 months of pasireotide.

Circulating adipokines were evaluated in patients with CD compared to a matched group of 12 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with active Cushing's disease.

Exclusion Criteria:

* pituitary radiotherapy treatment performed less than 5 years before pasireotide,
* pregnancy,
* women taking oral contraceptives,
* diabetes on GLP-1 analogues,
* DPP4 inhibitors or sulphonylureas treatment,
* intolerance to SSA,
* risk conditions for prolonged QT syndrome and severe liver o renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
Change of circulating adipokines levels | Change from baseline to 12 months of therapy
Change of homeostasis model assessment (HOMA-β ) | Change from baseline to 6 and 12 months of therapy
Change of area under the curve (AUC2h) of C-peptide during a mixed meal tolerance test | Change from baseline to 6 and 12 months of therapy
Change of M value evaluated by the euglycemic hyperinsulinemic clamp | Change from baseline to 12 months of therapy

IPD SHARING:
Plan to Share IPD: No